CLINICAL TRIAL: NCT01695993
Title: Alternative Approaches for Nausea Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Joseph Roscoe, Research Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UCCS1202; R01AT007474-01A1 (NIH)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Nausea
Keywords: Nausea; Quality of life; Chemotherapy; Expectancy
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Standard Care Only (No Intervention): Patients will receive standard care only
- Arm 2 - Expectancy-neutral Arm (Other): Patients receive:
  1. Expectancy-neutral handout
  2. Expectancy-neutral MP3
  3. Acupressure bands
  Interventions: Device: Acupressure bands; Other: Expectancy-neutral handout; Behavioral: Expectancy-neutral MP3
- Arm 3 - Expectancy-enhancing Arm (Experimental): Patients receive:
  1. Expectancy-enhancing handout
  2. Expectancy-enhancing MP3
  3. Acupressure bands
  Interventions: Device: Acupressure bands; Other: Expectancy-enhancing handout; Behavioral: Expectancy-enhancing MP3

INTERVENTIONS:
Device: Acupressure bands — Bilateral acupressure wrist bands
  Arms: Arm 2 - Expectancy-neutral Arm; Arm 3 - Expectancy-enhancing Arm
Other: Expectancy-neutral handout — The expectancy neutral handout has neutral information regarding the acupressure bands
  Arms: Arm 2 - Expectancy-neutral Arm
Behavioral: Expectancy-neutral MP3 — Patients will be given a portable MP3 player and relaxation MP3 that is about 12 minutes in length with a flute music background and guided imagery.
  Arms: Arm 2 - Expectancy-neutral Arm
Other: Expectancy-enhancing handout — The expectancy enhancing handout has expectancy-enhancing information regarding the acupressure bands
  Arms: Arm 3 - Expectancy-enhancing Arm
Behavioral: Expectancy-enhancing MP3 — Patients will be given a portable MP3 player and relaxation MP3 that is about 12 minutes in length with a flute music background and guided imagery. It also has expectancy-enhancing information regarding the acupressure bands.
  Arms: Arm 3 - Expectancy-enhancing Arm

SUMMARY:
216 Chemotherapy-naïve, female breast cancer patients about to begin chemotherapy and who expect to have nausea, will be entered. Participants will be randomized to one of three study arms: Arm 1: control; Arm 2: Expectancy-neutral handout + Expectancy-neutral MP3+ acupressure bands; Arm 3: Expectancy-enhancing handout + Expectancy-enhancing MP3 + acupressure bands.

Hypothesis: Acupressure bands provided with the relaxation MP3 will be effective in controlling chemotherapy-induced nausea

DETAILED DESCRIPTION:
Earlier research has shown that the effectiveness of acupressure bands in reducing nausea could be enhanced by boosting patients' expectations of the bands' efficacy. The present study seeks to confirm and extend these findings in a multi-site, 3-arm, randomized, controlled study of 216 breast cancer patients beginning chemotherapy who expect to have nausea. All patients will receive a standardized antiemetic regimen. Arm 1: control; Arm 2: Expectancy-neutral handout + Expectancy-neutral MP3+ acupressure bands; Arm 3: Expectancy-enhancing handout + Expectancy-enhancing MP3 + acupressure bands. The investigators hypothesize that acupressure bands provided with the relaxation MP3 will be effective in controlling chemotherapy-induced nausea. The two versions of the handout and MP3 are being examined to determine what is the most effective way to deliver the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be female.
* Have a diagnosis of breast cancer, any stage.
* Be chemotherapy naïve and about to begin her first course of chemotherapy.
* Be scheduled to receive one of the following four common chemotherapy regimens with the specified antiemetic regimen. They are:

  1. Chemotherapy regimen: Doxorubicin/cyclophosphamide. Antiemetic regimen: Aprepitant + palonosetron + dexamethasone on Day 1 and aprepitant + dexamethasone on Days 2 & 3.
  2. Chemotherapy regimen: Doxorubicin/cyclophosphamide/docetaxel. Antiemetic regimen: Aprepitant + palonosetron + dexamethasone on Day 1 and aprepitant + dexamethasone on Days 2 & 3.
  3. Chemotherapy regimen: Docetaxel/carboplatin. Antiemetic regimen: Palonosetron on Day 1 + dexamethasone on Days 1, 2, & 3.
  4. Chemotherapy regimen: Docetaxel/cyclophosphamide. Antiemetic regimen: Palonosetron on Day 1 + dexamethasone on Days 1, 2, & 3.

Note: Fosaprepitant will be allowed in place of aprepitant, and either granisetron or ondansetron, on one or more days, will be allowed in place of palonosetron.

* Have a response of > 3 or greater on a question assessing expected nausea as assessed on a 5-point Likert-scale anchored at one end by 1 = "I am certain I WILL NOT have this," and at the other end by 5 = "I am certain I WILL have this."
* Be able to read English (since the assessment materials are in printed format).
* Be 18 years of age or older and give written informed consent.

Exclusion Criteria:

* Have clinical evidence of lymphedema, current bowel obstruction, or symptomatic brain metastases, as determined by their treating oncologist.
* Be receiving concurrent radiotherapy or interferon.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Roscoe, Ph.D., Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Rochester General Hospital's Lipson Cancer and Blood Center, Rochester, New York
  - University of Rochester James P. Wilmot Cancer Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients receive standard care only
- Arm 2: Handout without expectancy- enhancing component Relaxation MP3 without expectancy-enhancing component
  - Acupressure bands
- Arm 3: Handout with expectancy- enhancing component Relaxation MP3 with expectancy- enhancing component Acupressure bands
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 81 | 80 | 81
Completed | 76 | 75 | 75
Not Completed | 5 | 5 | 6
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — To ill to continue | 1 | 2 | 0
Not completed — Changed Medical Facility | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Patients will receive only standard care
- Arm 2: * Handout without expectancy- enhancing component
  * Relaxation MP3 without expectancy-enhancing component
  * Acupressure bands
- Arm 3: * Handout with expectancy- enhancing component
  * Relaxation MP3 with expectancy-enhancing component
  * Acupressure bands
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 76 | 75 | 75 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.5) | 53.2 (11.6) | 52.6 (10.5) | 53 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 75 | 75 | 226
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 73 | 74 | 73 | 220
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 6 | 19
  White | 67 | 66 | 66 | 199
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 75 | 226

OUTCOME MEASURES:

1. Primary Outcome: Patient Report Nausea Diary
Description: Nausea and will be measured by a patient report diary completed by patients over a five-day period. Each day is divided into four segments (morning, afternoon, evening, night) in which patients report the severity of nausea and number of vomiting episodes for each period of the day. Severity of nausea is assessed on a 7-point rating scale, anchored at one end by 1 = "Not at all nauseated" and at the other end by 7 = "Extremely nauseated." The outcome variable for the primary analysis was greatest reported nausea from the five day period.
Time Frame: five days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Care: Patients receive only standard care
- Expectancy-Neutral Condition: * Handout without expectancy- enhancing component
  * Relaxation MP3 without expectancy-enhancing component
  * Acupressure bands
- Expectancy-Enhancing Condition: * Handout with expectancy-enhancing component
  * Relaxation MP3 with expectancy-enhancing component
  * Acupressure bands
Arm/Group | Standard Care | Expectancy-Neutral Condition | Expectancy-Enhancing Condition
Number analyzed (Participants) | 76 | 75 | 75
units on a scale | 3.87 (2.00) | 3.55 (2.00) | 3.52 (1.73)
Statistical Analysis 1: Comparison: Expectancy-Neutral Condition vs Expectancy-Enhancing Condition; Test type: Other — Primary Analysis: The Primary Aim to determine whether acupressure bands provided with efficacy-enhancing supplementary material are more effective in controlling chemotherapy-induced nausea than acupressure bands provided with neutral supplementary material was examined using ANCOVA with Peak Nausea after the first chemotherapy as the response, Arm (Arms 2 and 3) as the factor and expectancy of acupressure bands as the covariate; p = .05, ANCOVA — Not adjusted; Mean Difference (Net) = 0.03, Standard Deviation 1.9

ADVERSE EVENTS:
Time Frame: two months
Description: We used a standard definition for adverse events, but because this was a minimal risk study, our IRB required us to report and record only SAEs that were possibly, probably, or definitely related to the study intervention. See Section 5.7.1.1 of the protocol.
Groups:
- Arm 2: Patients receive:
  1. Handout without expectancy- enhancing component
  2. Relaxation MP3 without expectancy-enhancing component
  3. Acupressure bands
- Arm 3: Patients receive:
  1. Handout with expectancy- enhancing component
  2. Relaxation MP3 with expectancy-enhancing component
  3. Acupressure bands
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT01695993/Prot_SAP_000.pdf